CLINICAL TRIAL: NCT04700670
Title: Evaluation of the Effect of Dextran Sulphate on Anti-Xa Activities Measured in Patients Treated With Unfractionated Heparin in Different Indications-DEXHEP
Brief Title: Evaluation of the Effect of Dextran Sulphate on Anti-Xa Activities Measured
Acronym: DEXHEP
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC19_3001_DEXHEP
Record Dates: First submitted 2021-01-05; First posted 2021-01-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Unfractionated Heparin Treatment
Keywords: dextran sulphate; anti-Xa activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The measurement of anti-Xa activities will be carried out on frozen-defrosted plasma citrate and CTAD (Citrate-Theophylline, Adenosine, Dipyrioledam) with 4 reagents
  The dosage of platelet factor 4 and of the beta-TG will be carried out on frozen-defrosted plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: patients with cardiac surgery with CBP. Blood samples in the operating room, 5 to 10 minutes after neutralization of heparin by protamine
  Interventions: Biological: measurement of anti-Xa activities
- Group 2: patients who had cardiac surgery with CBP, between day 1 and day 5 after surgery.
  Interventions: Biological: measurement of anti-Xa activities
- Group 3: hospitalized patients in intensive care unit, including patients on extracorporeal life support (ECLS).
  Interventions: Biological: measurement of anti-Xa activities
- Group 4: patients hospitalized in a medical non-intensive care ward.
  Interventions: Biological: measurement of anti-Xa activities

INTERVENTIONS:
Biological: measurement of anti-Xa activities — The measurement of anti-Xa activities will be carried out on frozen-defrosted plasma citrate and CTAD with 4 reagents
  * STA-Liquid anti-Xa (STAGO) (not containing dextran)
  * Biophen Heparin LRT (Hyphen) (reactive containing dextran)
  * Berichrom (Siemens) with dextran
  * Berichrom (Siemens) without dextran
  The dosage of platelet factor 4 and of the beta-TG will be carried out on frozen-defrosted plasma with the asserachrom PF4 and Asserachrom beta-TG (Diagnostica Stago) kits.
  Other Names: dosage of platelet factor 4 and of the beta-TG

SUMMARY:
The measurement of anti-Xa activity is classically used for the dose adjustement of unfractionated heparin (UFH) treatment and to monitor reversal of UFH by protamine during cardiac surgery with cardiopulmonary bypass (CPB). Three categories of reagents are currently available in France for the measurement of anti-Xa activity: antithrombin-containing reagents (very little used), antithrombin-free reagents and antithrombin-free reagents with dextran sulphate. Significant differences in anti-Xa results based on the reagents used were described, particularly after protamine neutralization in CPB. Indeed, dextran sulphate, contained in some reagents, could dissociate the heparin/protamine complex contributing to the higher levels of anti-Xa with these reagents. The differences observed in these patients are likely related to the presence of platelet factor 4 (PF4) in the samples from either PF4 present in vivo in patients or released in vitro after blood collection. These differences may lead to different therapeutic attitudes, including the re-administration of protamine to neutralize heparin at the end of CBP

DETAILED DESCRIPTION:
Any hospitalized patient receiving UFH in the intensive, cardiac surgery and medicine departments of the participating centres will be offered the study by investigator. It will be included in the study after validation of the selection criteria and after collecting its non-opposition. This participation will not change the medical care of the participants.

Patients will be divided into four groups:

* Group 1: patients with cardiac surgery with CBP. Blood samples in the operating room, 5 to 10 minutes after neutralization of heparin by protamine.
* Group 2: patients who had cardiac surgery with CBP, between day 1 and day 5 after surgery.
* Group 3: hospitalized patients in intensive care unit, including patients on extracorporeal life support (ECLS).

Group 4: patients hospitalized in a medical non-intensive care ward.

The response to heparin treatment varies considerably depending on the clinical situation. The results found in one indication are not transposable to another indication. The 4 patient groups will provide a comprehensive response to situations in which heparin is used.

For each patient, during the usual follow-up of anti-Xa activity, and only once per patient, 3 to 4 additional blood tubes - 1 citrate tube (0.109 M) of 5 mL or 2 citrate tubes of 3 mL and 2 tubes CTAD (Citrate-Theophylline, Adenosine, Dipyrioledam) of 3 mL - will be taken during a blood test carried out in common practice. Thus, no additional invasive gestures are added by this search. CTAD contains, in addition to citrate, a platelet activation inhibitor and thus limits the in-vitro activation of platelets and thus the release of PF4.

Blood samples will be handle according to the usual procedures of each centre. All plasma will be aliquoted and stored at -80oC, until the end of inclusions in the hematology laboratories of each center.

At the end of the inclusion period, the aliquotes will be sent to the hematology laboratories of the Necker University Hospital and the University Hospital of Rennes for centralized testing.

The measurement of anti-Xa activities will be carried out on frozen-defrosted citrate and CTAD plasma with with 4 reagents:

* STA-Liquid anti-Xa (STAGO) (not containing dextran)
* Biophen Heparin LRT (Hyphen) (containing dextran)
* Berichrom (Siemens) with dextran
* Berichrom (Siemens) without dextran

The dosage of platelet factor 4 and beta-TG will be performed on frozen-defrosted plasma with CTAD with asserachrom PF4 and Asserachrom beta-TG (Diagnostica Stago) kits.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18;
* Hospitalized patients to receive UFH;
* No patient opposition.

Patients will be divided into four groups:

* Group 1: patients with cardiac surgery with CBP. Blood samples in the operating room, 5 to 10 minutes after neutralization of heparin by protamine.
* Group 2: patients who had cardiac surgery with CBP, between day 1 and day 5 after surgery.
* Group 3: hospitalized patients in intensive care unit, including patients on extracorporeal life support (ECLS).

Group 4: patients hospitalized in a medical non-intensive care ward..

Exclusion Criteria:

* pregnant or lactating women;
* adults subject to legal protection (safeguarding of justice, guardianship, guardianship), persons deprived of their liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any hospitalized patient receiving UFH in the intensive, cardiac surgery and medicine departments
Sampling Method: Non-Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2021-01-16 (Actual); Study Completion 2021-01-16 (Actual)

PRIMARY OUTCOMES:
Assess the effect of different reagents containing or not dextran sulphate, on the measurement of anti-Xa for different groups of patients | 5 days
  Measure of anti-Xa activity in CTAD plasma

SECONDARY OUTCOMES:
To define factors that influence the results of the biological test "anti-Xa" activity :type of anticoagulant (CTAD or citrate) . | 5 days
  Measure of anti-Xa activity
To define factors that influence the results of the biological test "anti-Xa" activity :concentration of platelet factor 4 (PF4) and beta-TG present in plasma | 5 days
  Measure of anti-Xa activity
To define factors that influence the results of the biological test "anti-Xa" activity :Patient characteristics including age and sex and if available, creatinine clearance, antithrombin, fibrinogen, platelet count | 5 days
  Measure of anti-Xa activity
To define factors that influence the results of the biological test "anti-Xa" activity :The indication of treatment | 5 days
  Measure of anti-Xa activity

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Gouin, Principal Investigator — Rennes University Hospital
Locations (8):
- France (8):
  - CHU Bordeaux, Bordeaux
  - CHU de Dijon, Dijon
  - CH de Versailles, Le Chesnay
  - CHU de Lille, Lille
  - APHP, CHU Lariboisière, Paris
  - APHP, HOPITAL Necker enfants malades, Paris
  - Rennes University Hospital, Rennes
  - CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lasne D, Toussaint-Hacquard M, Delassasseigne C, Bauters A, Flaujac C, Savard P, Mouton C, De Maistre E, Stepanian A, Eschwege V, Delrue M, Georges JL, Gros A, Mansour A, Leroy G, Jouffroy R, Mattei M, Beurton A, Pontis A, Neuwirth M, Nedelec-Gac F, Lecompte T, Curis E, Siguret V, Gouin-Thibault I. Factors Influencing Anti-Xa Assays: A Multicenter Prospective Study in Critically Ill and Noncritically Ill Patients Receiving Unfractionated Heparin. Thromb Haemost. 2023 Dec;123(12):1105-1115. doi: 10.1055/s-0043-1770096. Epub 2023 Jun 15. PMID 37321244